CLINICAL TRIAL: NCT00780104
Title: A Prospective Single Institution Pilot Study Evaluating the Pharmacokinetics of Sirolimus in Combination With MEC (Mitoxantrone + Etoposide + Cytarabine) in Patients With High Risk Leukemias
Brief Title: Sirolimus in Combination With MEC in High Risk Myeloid Leukemias
Acronym: UPCC 02407
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02407
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Myeloid Leukemias; AML; Leukemia; CML
Keywords: Advanced myeloid leukemias; AML; Leukemia; Relapsed myeloid leukemias; Refractory myeloid leukemias; MEC; Rapamycin; Sirolimus
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia | interventions — Sirolimus; Mitoxantrone; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapamycin + MEC (Experimental)
  Interventions: Drug: Rapamycin, Mitoxantrone, Etoposide, Cytarabine; Drug: Rapamycin + MEC

INTERVENTIONS:
Drug: Rapamycin, Mitoxantrone, Etoposide, Cytarabine — Rapamycin loading dose of 12 mg followed by a single daily dose for 8 days of 4 mg/day + MEC (Mitoxantrone 8 mg/m2/day IV, Etoposide 100 mg/m2/day IV and Cytarabine 1000 mg/m2 IV every 24 hours for 5 days. Starts after 4th dose of sirolimus.
Drug: Rapamycin + MEC — Rapamycin loading dose of 12 mg followed by a single daily dose for 8 days of 4 mg/day + MEC (Mitoxantrone 8 mg/m2/day IV, Etoposide 100 mg/m2/day IV and Cytarabine 1000 mg/m2 IV every 24 hours for 5 days. Starts after 4th dose of sirolimus.

SUMMARY:
The purpose of this study is to evaluate the side effects of sirolimus (rapamycin) given in combination with chemotherapy (Mitoxantrone + Etoposide + Cytarabine (MEC)) on high risk myeloid leukemias.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologic evidence of advanced myeloid leukemias defined as one of the following: primary refractory non-M3 AML; relapsed non-M3 AML; secondary AML; intermediate or poor prognosis de novo AML in patients who are >= 60 years old
* >= 18 years of age
* ECOG performance status of 0, 1
* Able to consume oral medication
* Initial laboratory values: creatinine <= 2.0 mg/dL; total or direct bilirubin <= 1.5/dL; SGPT(ALT) <= 3xULN; negative pregnancy test for women with child-bearing potential
* Ejection fraction of >= 45%

Exclusion Criteria:

* Subjects with FAM B3
* Must not be receiving chemotherapy (except Hydroxyurea)
* Not receiving growth factors, except for erythropoietin
* Subjects with a "currently active" second malignancy other than non-melanoma skin cancers
* Subjects with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, MI within the last 6 months or uncontrolled cardiac arrhythmia
* Subjects taking diltiazem
* Subjects who require HIV protease inhibitors or those with AIDS-related illnesses
* No evidence of cerebellar dysfunction at baseline or during prior cytarabine therapy
* Not pregnant or breastfeeding
* Uncontrolled infection
* Subjects taking Carbamazepine, Rifabutin, Rifampin, Rifapentine, St. John's wort, Clarithromycin, Cyclosporine, Diltiazem, Erythromycin, Telithromycin, Verapamil, Tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assessment of biologic effects of rapamycin on mTOR targets such as p70 protein phosphorylation in leukemic cells | Study conclusion

SECONDARY OUTCOMES:
Safety of the sirolimus + MEC regimen | Study conclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania, United States